CLINICAL TRIAL: NCT05731973
Title: Intercostal Nerve Cryoablation Versus Thoracic Epidural Analgesia for Minimal Invasive Nuss Repair of Pectus Excavatum: a Randomized Clinical Trial (ICE Trial)
Brief Title: Intercostal Nerve Cryoablation Versus Epidural Analgesia for Nuss Repair of Pectus Excavatum
Acronym: ICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: AtriCure, Inc. (Industry)
Responsible Party: Principal Investigator, Erik de Loos, Principal investigator, Zuyderland Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Z2023005
Record Dates: First submitted 2023-01-26; First posted 2023-02-16 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Pectus Excavatum; Funnel Chest
Keywords: Pectus Excavatum; Funnel Chest; Intercostal nerve cryoablation; Analgesia
MeSH Terms: conditions — Funnel Chest; Agnosia | interventions — Cryosurgery; Tea; Sufentanil; Bupivacaine; Injections, Epidural; Analgesics, Opioid; Oxycodone; Health Services Needs and Demand

STUDY DESIGN:
Intervention Model Description: Single center, prospective, unblinded, randomized clinical trial. Block randomization, including stratification based on age (12-16 years and 17-24 years) and sex, with an allocation ratio of 1:1 will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercostal nerve cryoablation (Experimental): When a patient is allocated to the intercostal nerve cryoablation group, cryoablation will be performed prior to bar placement. In brief, cryoablation will be performed at the level of the bar and two levels above and below, bilaterally. For this, a second portal access will be placed for video guidance on the contralateral side, and the cryoprobe (cryoICE, Atricure, Masion, OH, USA) will be inserted through the thoracic incisions that are already made for bar placement. The probe will be placed at the inferior aspect of the ribs, posterior to the midaxillary line, directly on the neurovascular bundle. One freezing cycle takes 2 minutes, and a temperature of -60 ⁰C will be applied. The probe will be warmed to room temperature before removing it from the pleura to prevent additional trauma. Furthermore, intercostal nerve cryoablation will be combined with single shot bupivacaine (1.25 mg/ml) intercostal nerve blocks placed just anterior to the side of the cryoablation.
  Interventions: Procedure: Intercostal nerve cryoablation; Drug: Intercostal nerve block (single shot bupivacaine (1.25 mg/ml)); Drug: Opioids (oxycodone with prolonged discharge 10 mg PO every 12 hours and oxycodone 5 mg every 6 hours, as needed)
- Thoracic epidural (local continuous infusion with sufentanyl (1 µg/ml) and bupivacaine (1.25 mg/ml)) (Active Comparator): Prior to surgery, an anesthesiologist will place the thoracic epidural at T5-T6 or T6-T7 interspace in the awake patient. After correct placement, a local continuous infusion with sufentanyl (1 µg/ml) and bupivacaine (1.25 mg/ml) will be started. At the third postoperative day, thoracic epidural analgesia will be ceased and transitioned to oral pain medication at discretion of the pain management team. In general, opioids (oxycodone with prolonged discharge 10 mg PO every 12 hours and oxycodone 5 mg every 6 hours as needed) will be provided 12 hours before thoracic epidural analgesia is ceased.
  Interventions: Drug: Thoracic epidural analgesia (continuous infusion with sufentanyl (1 µg/ml) and bupivacaine (1.25 mg/ml)); Drug: Opioids (oxycodone with prolonged discharge 10 mg PO every 12 hours and oxycodone 5 mg every 6 hours, as needed)

INTERVENTIONS:
Procedure: Intercostal nerve cryoablation — Intercostal nerve cryoablation is applied during Nuss procedure.
  Other Names: Cryoablation
  Arms: Intercostal nerve cryoablation
Drug: Thoracic epidural analgesia (continuous infusion with sufentanyl (1 µg/ml) and bupivacaine (1.25 mg/ml)) — Thoracic epidural is placed prior to Nuss procedure
  Other Names: Epidural
  Arms: Thoracic epidural (local continuous infusion with sufentanyl (1 µg/ml) and bupivacaine (1.25 mg/ml))
Drug: Intercostal nerve block (single shot bupivacaine (1.25 mg/ml)) — Single shot bupivacaine (1.25 mg/ml) intercostal nerve blocks are placed just anterior to the side of the cryoablation.
  Other Names: Intercostal nerve block
  Arms: Intercostal nerve cryoablation
Drug: Opioids (oxycodone with prolonged discharge 10 mg PO every 12 hours and oxycodone 5 mg every 6 hours, as needed) — Opioids
  Other Names: opioids, oxycodone (with prolonged discharge)

SUMMARY:
Primary objective of the current study is to determine the impact of intercostal nerve cryoablation on postoperative length of hospital stay compared to standard pain management of young pectus excavatum patients (12-24 years) treated with the minimal invasive Nuss procedure. The study is designed as a single center, prospective, unblinded, randomized clinical trial.

DETAILED DESCRIPTION:
Rationale: The minimal invasive Nuss procedure is currently considered the treatment of choice for pectus excavatum. This procedure is usually associated with severe postoperative pain as great forces are employed on the thoracic cage to correct the sternal depression. Pain is the main limiting factor for early discharge. Epidural analgesia is currently considered gold standard for postoperative pain treatment. Alternative pain management strategies (e.g., patient-controlled analgesia and paravertebral nerve block) have also been described but fail in accomplishing adequate prolonged post-operative pain management. Alternatively, continuous use of opioids comes with side-effects like severe nausea, urinary retention and obstipation. Intercostal nerve cryoablation seems a promising novel technique for postoperative analgesia. Prior studies comparing intercostal cryoablation to other pain treatment modalities after pectus excavatum repair through the minimal invasive Nuss procedure report promising results, but pose significant limitations (e.g., small sample size, retrospective nature with non-matched patient groups or considerable confounders).

Objective: Primary objective of the current study is to determine the impact of intercostal nerve cryoablation on postoperative length of hospital stay compared to standard pain management of young pectus excavatum patients treated with the minimal invasive Nuss procedure.

Study design: The study protocol is designed for a single center, prospective, unblinded, randomized clinical trial.

Study population & intervention: Intercostal nerve cryoablation will be compared to thoracic epidural analgesia in young pectus excavatum patients (i.e., 12-24 years of age) treated with the minimal invasive Nuss procedure. Block randomization, including stratification based on age (12-16 years and 17-24 years) and sex, with an allocation ratio of 1:1 will be performed.

Main study parameters/endpoints: Postoperative length of hospital stay will be recorded as the primary endpoint. Secondary outcomes include: 1) pain intensity; 2) operative time; 3) opioid usage; 4) complications, including neuropathic pain; 5) creatine kinase activity; 6)intensive care unit admissions; 7) readmissions; 8) postoperative mobility; 9) health related quality of Life; 10) days to return to work/school; 11) number of postoperative outpatient visits and 12) hospital costs.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risks for study participants are negligible as the cryoablation technique has already been effectively used in the Nuss procedure without any serious side effects. Also, participants will be monitored daily by nursing staff and surgeons while admitted to the hospital. Burden associated with participation in the current study consists of completion of several questionnaires preoperatively and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing the minimal invasive Nuss procedure for surgical repair of pectus excavatum.
* Young patients (12-24 years of age) according to the definition used by the World Health Organization. This cut-off point is chosen to create a more homogenous patient sample, as the thoracic cage is fully matured by the age of 24, in size and density, which will have an effect on postoperative pain.

Exclusion Criteria:

* A chest wall deformity other than pectus excavatum;
* Opioid use in the 3 months prior to surgery;
* Pain syndrome (e.g., fibromyalgia) or neuropathic pain prior to surgical repair of pectus excavatum;
* Connective tissue disease (e.g., Marfan syndrome, Ehlers-Danlos syndrome);
* Previous thoracic surgery or pectus excavatum repair;
* Contraindication for intercostal nerve cryoablation or thoracic epidural analgesia (e.g., patient refusal, infection at the site of cannulation, uncontrolled systemic infection, bleeding diathesis, increased intracranial pressure, mechanical spine obstruction);
* Psychiatric disease currently receiving treatment;
* Not mastering the Dutch language;
* Participation in another clinical trial that may interfere with the current trial.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Hospitalization period, average of 5 days
  Number of days of hospital admittance after the Nuss procedure.

SECONDARY OUTCOMES:
Pain intensity | Preoperative care unit before surgery, in the morning on postoperative day 1 and 2, and 7 days, 14 days, 3 months and 6 months post operation
  Pain intensity at rest and during mobilization. Pain scores will be rated on the numeric rating scale (NRS, 1-10)
Operative time | During Nuss procedure
  Operative time in minutes. Duration of cryoablation will be assessed separately. Operative time will not include the time needed for the placement of the thoracic epidural as placement will be performed in the preoperative care unit.
Opioid usage | postoperative day 1 and 2, and first 2 weeks after surgery
  A) Intraoperative administered opioids; B) Opioid usage during postoperative day 0, 1 and 2 at the recovery unit and surgical ward; C) Opioid usage within the first 2 weeks after surgery. Opioid usage will be converted to oral morphine milligram equivalents (MME).
Complications | 6 months postoperative
  Complications graded according to the Clavien-Dindo classification. The most common procedure- and analgesia-related complications are defined in Supplementary Materials Table 1-2 for transparency, including neuropathic pain. Occurrence of neuropathic pain will be actively monitored during the hospitalization period, and during all follow-up appointments.
Creatine kinase (CK) activity | Preoperative and day 1 postoperative
  CK levels will be assessed prior to the surgical procedure (i.e., baseline measurement during routine blood evaluation on the day of surgery) and on postoperative day 1. CK levels will be denoted in U/L.
Intensive care unit admission | Hospitalization period, average of 5 days
  Intensive care unit admission due to the occurrence of perioperative complications in absolute numbers
Length of intensive care unit admission | Hospitalization period, average of 5 days
  Length of admission due to the occurrence of perioperative complications in absolute numbers.
Number of readmissions | 6 months postoperative
  Number of readmissions denoted as absolute numbers.
Length of readmissions | 6 months postoperative
  length of readmissions denoted as absolute numbers.
Degree of mobility | Postoperative day 1 and 2
  Degree of mobility measured on a 4-point scale (i.e., 1. on the bed, 2. to the chair, 3. to the toilet, 4. outside the patient's hospital room) during postoperative day 1 and 2.
HRQOL - PEEQ | Before surgery as a baseline measurement, and at 2 weeks, 3 months and 6 months after the surgical procedure
  HRQOL, measured by the Dutch version of the pectus evaluation questionnaire (PEEQ). The PEEQ is a validated disease specific questionnaire evaluating the quality of life in pectus excavatum patients (37,38).
HRQOL - SF-36 | Before surgery as a baseline measurement, and at 2 weeks, 3 months and 6 months after the surgical procedure
  HRQOL, measured by the Dutch version of the short form health survey (SF-36)(37-40). The SF-36 is a generic questionnaire that taps health in eight dimensions (39).
HRQOL - EQ-5D-5L | Before surgery as a baseline measurement, and at 2 weeks, 3 months and 6 months after the surgical procedure
  HRQOL, measured by the Dutch version of the EuroQol 5 dimensions 5 levels (EQ-5D-5L) (37-40). For the EQ-5D-5L, participants will rate their health in 5 dimensions on 5 levels and will give an overall score of their health on a visual analogue scale (VAS) (40).
Days to return to work/school | 6 months postoperative
  Days to return to work/school, reported as days between discharge from hospital and return to work or school.
Postoperative visits | 6 months postoperative
  Number of postoperative outpatient visits and telephone appointments denoted as absolute numbers in the first 6 months after the surgical procedure.
Hospital costs | 6 months postoperative
  Hospital costs, reported as hospital costs during initial hospitalization (e.g., medication, patient care supply, surgical equipment), and hospital costs after discharge until 6 months follow-up (e.g., medications, outpatient visits, (opioid related) readmissions).

CONTACTS AND LOCATIONS:
Overall Officials: Erik R De Loos, Principal Investigator — Zuyderland Medical Center
Locations (1):
- Zuyderland Medical Center, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Croitoru DP, Kelly RE Jr, Goretsky MJ, Lawson ML, Swoveland B, Nuss D. Experience and modification update for the minimally invasive Nuss technique for pectus excavatum repair in 303 patients. J Pediatr Surg. 2002 Mar;37(3):437-45. doi: 10.1053/jpsu.2002.30851. PMID 11877663
- [Result] Nuss D. Minimally invasive surgical repair of pectus excavatum. Semin Pediatr Surg. 2008 Aug;17(3):209-17. doi: 10.1053/j.sempedsurg.2008.03.003. PMID 18582827
- [Result] Nuss D, Kelly RE Jr. Indications and technique of Nuss procedure for pectus excavatum. Thorac Surg Clin. 2010 Nov;20(4):583-97. doi: 10.1016/j.thorsurg.2010.07.002. PMID 20974443
- [Result] Dekonenko C, Dorman RM, Duran Y, Juang D, Aguayo P, Fraser JD, Oyetunji TA, Snyder CL, Holcomb GW 3rd, Millspaugh DL, St Peter SD. Postoperative pain control modalities for pectus excavatum repair: A prospective observational study of cryoablation compared to results of a randomized trial of epidural vs patient-controlled analgesia. J Pediatr Surg. 2020 Aug;55(8):1444-1447. doi: 10.1016/j.jpedsurg.2019.09.021. Epub 2019 Oct 26. PMID 31699436
- [Result] Qi J, Du B, Gurnaney H, Lu P, Zuo Y. A prospective randomized observer-blinded study to assess postoperative analgesia provided by an ultrasound-guided bilateral thoracic paravertebral block for children undergoing the Nuss procedure. Reg Anesth Pain Med. 2014 May-Jun;39(3):208-13. doi: 10.1097/AAP.0000000000000071. PMID 24682079
- [Result] Sertcakacilar G, Kose S. Bilateral PECS II Block is Associated with Decreased Opioid Consumption and Reduced Pain Scores for up to 24 hours After Minimally Invasive Repair of Pectus Excavatum (Nuss Procedure): A Retrospective Analysis. J Cardiothorac Vasc Anesth. 2022 Oct;36(10):3833-3840. doi: 10.1053/j.jvca.2022.06.001. Epub 2022 Jun 6. PMID 35817669
- [Result] Abdel Shaheed C, McLachlan AJ, Maher CG. Rethinking "long term" opioid therapy. BMJ. 2019 Nov 29;367:l6691. doi: 10.1136/bmj.l6691. No abstract available. PMID 31784472
- [Result] Cadaval Gallardo C, Martinez J, Bellia-Munzon G, Nazar M, Sanjurjo D, Toselli L, Martinez-Ferro M. Thoracoscopic cryoanalgesia: A new strategy for postoperative pain control in minimally invasive pectus excavatum repair. Cir Pediatr. 2020 Jan 20;33(1):11-15. English, Spanish. PMID 32166917
- [Result] Aiken TJ, Stahl CC, Lemaster D, Casias TW, Walker BJ, Nichol PF, Leys CM, Abbott DE, Brinkman AS. Intercostal nerve cryoablation is associated with lower hospital cost during minimally invasive Nuss procedure for pectus excavatum. J Pediatr Surg. 2021 Oct;56(10):1841-1845. doi: 10.1016/j.jpedsurg.2020.10.009. Epub 2020 Oct 19. PMID 33199059
- [Result] Morikawa N, Laferriere N, Koo S, Johnson S, Woo R, Puapong D. Cryoanalgesia in Patients Undergoing Nuss Repair of Pectus Excavatum: Technique Modification and Early Results. J Laparoendosc Adv Surg Tech A. 2018 Sep;28(9):1148-1151. doi: 10.1089/lap.2017.0665. Epub 2018 Apr 19. PMID 29672193
- [Result] Harbaugh CM, Johnson KN, Kein CE, Jarboe MD, Hirschl RB, Geiger JD, Gadepalli SK. Comparing outcomes with thoracic epidural and intercostal nerve cryoablation after Nuss procedure. J Surg Res. 2018 Nov;231:217-223. doi: 10.1016/j.jss.2018.05.048. Epub 2018 Jun 21. PMID 30278932
- [Result] Sun RC, Mehl SC, Anbarasu CR, Portuondo JI, Espinoza AF, Whitlock R, Mazziotti MV. Intercostal cryoablation during Nuss procedure: A large volume single surgeon's experience and outcomes. J Pediatr Surg. 2021 Dec;56(12):2229-2234. doi: 10.1016/j.jpedsurg.2021.03.006. Epub 2021 Mar 17. PMID 33853732
- [Result] Sujka J, Benedict LA, Fraser JD, Aguayo P, Millspaugh DL, St Peter SD. Outcomes Using Cryoablation for Postoperative Pain Control in Children Following Minimally Invasive Pectus Excavatum Repair. J Laparoendosc Adv Surg Tech A. 2018 Nov;28(11):1383-1386. doi: 10.1089/lap.2018.0111. Epub 2018 Jun 21. PMID 29927703
- [Result] Daemen JHT, de Loos ER, Vissers YLJ, Bakens MJAM, Maessen JG, Hulsewe KWE. Intercostal nerve cryoablation versus thoracic epidural for postoperative analgesia following pectus excavatum repair: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2020 Oct 1;31(4):486-498. doi: 10.1093/icvts/ivaa151. PMID 32929487
- [Result] Graves CE, Moyer J, Zobel MJ, Mora R, Smith D, O'Day M, Padilla BE. Intraoperative intercostal nerve cryoablation During the Nuss procedure reduces length of stay and opioid requirement: A randomized clinical trial. J Pediatr Surg. 2019 Nov;54(11):2250-2256. doi: 10.1016/j.jpedsurg.2019.02.057. Epub 2019 Mar 17. PMID 30935731
- [Result] Zobel MJ, Ewbank C, Mora R, Idowu O, Kim S, Padilla BE. The incidence of neuropathic pain after intercostal cryoablation during the Nuss procedure. Pediatr Surg Int. 2020 Mar;36(3):317-324. doi: 10.1007/s00383-019-04602-1. Epub 2019 Nov 23. PMID 31760443
- [Derived] Janssen N, Daemen JHT, Franssen AJPM, van Polen EJ, van Roozendaal LM, Hulsewe KWE, Vissers Y, de Loos ER. Intercostal nerve cryoablation versus thoracic epidural analgesia for minimal invasive Nuss repair of pectus excavatum: a protocol for a randomised clinical trial (ICE trial). BMJ Open. 2024 Mar 25;14(3):e081392. doi: 10.1136/bmjopen-2023-081392. PMID 38531584
- See also: FDA — https://www.atricure.com/sites/default/files/pdf-doc/K200697.Letter.SE_.FINAL_Sent001.pdf